CLINICAL TRIAL: NCT01068795
Title: Dose Adjusting Enoxaparin Thromboprophylaxis Dosage According to Anti-factor Xa Plasma Levels Improve Pregnancy Outcome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Principal Investigator, Raed Salim, MD, HaEmek Medical Center, Israel
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 0048-09-EMC ANTIXA-02; 0048-09-EMC
Record Dates: First submitted 2010-01-20; First posted 2010-02-15 (Estimated); Last update posted 2016-02-23 (Estimated); Status verified 2016-02

CONDITIONS: Fetal Demise; Fetal Growth Restriction; Preeclampsia; Abruptio Placentae; Thromboembolism
Keywords: placental syndrome; maternal thromboembolic event; enoxaparin; anti-factor Xa
MeSH Terms: conditions — Fetal Death; Fetal Growth Retardation; Pre-Eclampsia; Abruptio Placentae; Thromboembolism | interventions — Enoxaparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- enoxaparin fixed (No Intervention): enoxaparin dosage will be fixed during pregnancy
- enoxaparin adjusted (Experimental): enoxaparin dosage will be adjusted according to anti-factor Xa plasma levels
  Interventions: Drug: enoxaparin

INTERVENTIONS:
Drug: enoxaparin — enoxaparin dosage will be adjusted according to anti-factor Xa plasma levels
  Arms: enoxaparin adjusted

SUMMARY:
The risk of venous thromboembolism increases in pregnancy. Thrombophilia whether genetic or acquired, is a hypercoagulable disorder that may increase the risk of venous thromboembolic events. Clinically, these events are presented as maternal deep vein thrombosis and pulmonary emboli. Thrombophilias are also associated with adverse fetal outcomes including intrauterine growth restriction, intrauterine fetal death, severe preeclampsia, placental abruption and recurrent abortions.

Pregnant women who experienced one or more of the above complications are advised to be examined for the presence of the genetic or the acquired form of thrombophilia.

Low molecular weight heparin prophylaxis, an anticoagulant, is advised for pregnant women with a history of thromboembolism, and many experts recommend prophylaxis for pregnant patients with a known thrombophilia and history of adverse pregnancy outcomes associated with these hypercoagulable states.

Physiologic changes in normal pregnancy, including weight gain, increased renal clearance and volume of distribution, may decrease the availability of low molecular weight heparin (Enoxaparin or Dalteparin), or produce a less predictable response in pregnant women compared with nonpregnant women. There are no clear recommendations for use of prophylactic low molecular weight heparin in pregnancy. Clinicians tend to use doses suggested for nonpregnant patients. Regarding pregnant patients taking enoxaparin or dalteparin, the American College of Obstetricians and Gynecologists states that "because of the lack of data regarding adequate dosing during pregnancy, anti-factor Xa levels may be monitored".

Two recently published studies demonstrated that plasma anti-factor Xa levels during pregnancy were lower than expected, indicating that many pregnant patients may receive a subprophylactic dosing.

Our objective is to check pregnancy outcome among thrombophilic women treated with an adjusted enoxaparin thromboprophylaxis dosage according to anti-factor Xa plasma levels compared to women with fixed dosage.

ELIGIBILITY:
Inclusion Criteria:

WOMEN WITH

* Singleton gestation
* A history of fetal demise, fetal growth restriction, placental abruption, preeclampsia, recurrent abortions or maternal thromboembolic event.
* Acquired or congenital thrombophilia treated with low molecular weight heparin

Exclusion Criteria:

* Women treated empirically with low molecular weight heparin
* Women with a history of pregestational diabetes.
* Significant polyhydramnios or oligohydramnios, major fetal structural, generic or chromosomal malformations

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 144 (Actual)
Dates: Start 2009-07; Primary Completion 2015-01 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
placental syndrome or thromboembolic event | 9 months

SECONDARY OUTCOMES:
enoxaparin side effects | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Raed Salim, MD, Principal Investigator — Dep. OB/GYN, HaEmek Medical Center, Afula, Israel
Locations (1):
- Dep. OB/GYN, HaEmek Medical Center, Afula, Israel

REFERENCES:
- [Derived] Middleton P, Shepherd E, Gomersall JC. Venous thromboembolism prophylaxis for women at risk during pregnancy and the early postnatal period. Cochrane Database Syst Rev. 2021 Mar 29;3(3):CD001689. doi: 10.1002/14651858.CD001689.pub4. PMID 33779986
- [Derived] Salim R, Nachum Z, Gavish I, Romano S, Braverman M, Garmi G. Adjusting enoxaparin dosage according to anti-FXa levels and pregnancy outcome in thrombophilic women. A randomised controlled trial. Thromb Haemost. 2016 Sep 27;116(4):687-95. doi: 10.1160/TH16-03-0221. Epub 2016 Jul 21. PMID 27440463